CLINICAL TRIAL: NCT00003758
Title: Treatment of Relapsed Acute Myelogenous Leukemia Consisting of Intermediate Dose Cytosine Arabinoside (ARA-C) Plus Interspaced Continuous Infusion Idarubicin, Followed by Continuous Infusion of Low-Dose ARA-C, A Phase II Study by the EORTC-LCG
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed Acute Myelogenous Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066882; EORTC-06956
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2001-01

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; adult acute monoblastic leukemia and acute monocytic leukemia (M5); childhood acute monoblastic leukemia and acute monocytic leukemia (M5); adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute erythroleukemia (M6); childhood acute eosinophilic leukemia; childhood acute basophilic leukemia; childhood acute megakaryocytic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Cytarabine; Idarubicin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: cytarabine
Drug: idarubicin
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of cytarabine plus idarubicin in treating patients who have relapsed acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility and efficacy of intermediate dose cytarabine plus idarubicin followed by low dose cytarabine in patients with relapsed acute myelogenous leukemia.

OUTLINE: This is a multicenter study. Patients receive intermediate dose cytarabine IV over 2 hours twice a day on days 1-5, idarubicin IV over 24 hours on days 1, 3, and 5, and low dose cytarabine IV over 24 hours on days 6-15. If patients achieve complete remission by day 35, this regimen is repeated once. If patients achieve partial remission by day 35, this regimen is repeated, except with an additional day of idarubicin on day 7. If these patients then achieve complete remission by day 70, the regimen is repeated. Patients may then undergo stem cell transplantation within 6 months of achieving complete remission. Patients who have an HLA identical sibling available receive an allogeneic transplant; others receive an autologous transplant. Patients are followed monthly for 1 year, every 3 months for 3 years, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 24-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: First bone marrow relapse of primary acute myelogenous leukemia (AML), all subtypes except M3 OR First bone marrow relapse of secondary AML that occurred after other malignancies, but cured, or after alkylating agents and/or radiotherapy, or after myelodysplastic syndrome No previously untreated AML or second or subsequent relapse of AML No isolated extramedullar localization of AML Must have achieved a first complete remission No leukemias after other myeloproliferative diseases

PATIENT CHARACTERISTICS: Age: 15 to 60 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 1.5 times ULN AST no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No cardiac contraindications to anthracycline chemotherapy Ventricular ejection fraction at least 45% Other: No uncontrolled infection No concurrent severe neurological or psychiatric disease No other progressive malignant nonhematological disease

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior allogeneic or autologous bone marrow or peripheral stem cell transplant Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Petra Muus, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (16):
- Belgium (4):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- Croatia (2):
  - Medical School/University of Zagreb, Zagreb
  - University Hospital Rebro, Zagreb
- France (2):
  - Hotel Dieu de Paris, Paris
  - Hopital Necker, Paris
- Italy (2):
  - Ospedale San Eugenio, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Netherlands (4):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Sint Joseph Ziekenhuis, Veldhoven
- Hospital Escolar San Joao, Porto, Portugal
- Ibn-i Sina Hospital, Ankara Univeristy, Ankara, Turkey (Türkiye)